CLINICAL TRIAL: NCT03596398
Title: Epidemiological Study of Fabry Disease in Taiwan Young Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chiayi Christian Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: 105028
Record Dates: First submitted 2018-06-15; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Fabry Disease
Keywords: Fabry disease; Young stroke
MeSH Terms: conditions — Fabry Disease | interventions — alpha-Galactosidase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Dried blood spot (DBS) sample and whole blood sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young stroke: Patients with acute stroke aged 20 or over, and under 56 years old (Not included 56) .
  Interventions: Genetic: GLA gene

INTERVENTIONS:
Genetic: GLA gene — Genetic test will be performed when enzyme activity is found abnormal in the whole blood test or confirmation is required. 5 ml of blood sample will be obtained and polymerase chain reaction (PCR) sequencing will be executed to determine mutations in the GLA gene.

SUMMARY:
Epidemiological Study of Fabry Disease in Taiwan Young Stroke Patients

DETAILED DESCRIPTION:
This is a cross-sectional, population-based study. No randomization procedure will be executed in this study. Approximately 1000 subjects over a 36-month period. The aim of this screening study is to identify the Fabry disease as the cause in patients with young stroke.

To measure the level of α-Gal A activity, male subjects will initially provide a DBS sample and female subjects will start with a test by whole blood sample.

The prevalence of Fabry disease among patients with young stroke will be estimated by a confirmative diagnosis in gene testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 or over
* Patients aged under 56 years old, not included 56
* Patients with acute stroke
* Patients and/or their legal representatives are willing to provide written informed consent

Exclusion Criteria:

* Patients with a confirmed diagnosis of Fabry disease

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young stroke
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Fabry disease | 3 years later
  The prevalence of Fabry disease in patients with young stroke